CLINICAL TRIAL: NCT02672579
Title: Study of Kids Itch Severity (SKIS): "Validation and Mobilization of Pediatric Pruritus Outcome Instruments"
Brief Title: Study of Kids Itch Severity (SKIS)
Acronym: SKIS
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suephy Chen, MD, Associate Professor, Emory University
Other Study IDs: IRB00081076
Record Dates: First submitted 2015-12-15; First posted 2016-02-03 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Chronic Pruritus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Children 4-7 years: Pediatric subjects between the ages of 4 and 7 who have had pruritus for 6 weeks or longer will complete surveys to assess the severity of pruritus.
- Children 8-17 years: Pediatric subjects between the ages of 8 and 17 who have had pruritus for 6 weeks or longer will complete surveys to assess the severity of pruritus.
- Parents: Parents of pediatric subjects between the ages of 4-17 years with chronic pruritus (for 6 weeks or longer) will complete surveys to assess their perception of their child's severity of pruritus.
- Clinicians: Clinicians treating pediatric subjects between the ages of 4-17 years with chronic pruritus (for 6 weeks or longer) will complete surveys to assess their perception of the child's severity of pruritus.

SUMMARY:
This purpose of this study is to validate two measures of chronic itching in kids: itch severity (ItchyQuant) and the impact on their quality of life (ItchyQoL).

DETAILED DESCRIPTION:
There are many diseases that affect children where the primary symptom is pruritus. This study aims to validate an age appropriate pediatric version of the ItchyQoL, a pruritus-specific quality of life instrument, and the ItchyQuant, a self-reported itch severity scale, to better understand how pruritus affects the pediatric population. These instruments will comprehensively capture the severity and impact of pruritus in children. The physicians want to explore the opportunity to integrate patient-reported outcome measures (PROM) as a patient-reported tool in the ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients between the ages of 4 and 17 (parents and clinicians will be older than 18 years, both male and female)
* Informed consent/assent signed and dated by the patient/parent
* Willingness and ability for the patient to commit to all follow-up visits/phone calls for the duration of the study

Exclusion Criteria:

* Inability to speak or read English
* Any other disabilities that would prevent them from completing a survey
* Unwillingness or inability for the patient to commit to all follow-up visits/phone calls for the duration of the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of 4 and 17 who have chronic pruritus (for 6 weeks or longer). The information detailed below is reflective of the pediatric population which is the primary focus of this study though the parents and clinicians will also complete surveys.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
ItchyQoL (TotsItchyQoL) test-retest reliability | Baseline
  Subjects in the 4-7 year age group will complete the TotsItchyQoL® questionnaire. This questionnaire has a total of 16 items with cartoons accompanying each question. The interviewer will ask the subjects questions to rate how pruritus affected their quality of life (QOL). The test-retest reliability will be assessed by analyzing the recorded responses to assess improvement, no change, or worsening of their pruritus.
ItchyQoL (KidsItchyQoL) test-retest reliability | Baseline
  Subjects in the 8-17 year age group will complete the KidsItchyQoL® questionnaire. This is a 27-item questionnaire where the subjects are asked to rate how pruritus affected their quality of life (QOL). The test-retest reliability will be assessed by analyzing the recorded responses to assess improvement, no change, or worsening of their pruritus.
ItchyQoL (TotsItchyQoL) validity | Baseline
  Subjects in the 4-7 year age group will complete the TotsItchyQoL® questionnaire. There are a total of 16 items with cartoons accompanying each question. The subjects will be asked to rate the severity of their pruritus and the responses will be recorded. Each response will be scored and the scores will be compared across pruritus severity; mild,moderate or severe; to assess the validity of the questionnaire.
ItchyQoL (KidsItchyQoL) validity | Baseline
  Subjects in the 8-17 year age group will complete the TotsItchyQoL® questionnaire. There are a total of 16 items with cartoons accompanying each question. The subjects will be asked to rate the severity of their pruritus and the responses will be recorded. Each response will be scored and the scores will be compared across pruritus severity; mild,moderate or severe; to assess the validity of the questionnaire.
Psychometric properties of the ItchyQuant | Baseline
  Age-appropriate ItchyQuant will be administered as follows; subjects 4-5 years will use the modified 3-point ItchyQuant, for subjects 6-7 years, the 3-point and 5-point ItchyQuant and for ages 8 and older, the traditional non-cartoon version of the numeric rating scale (NRS) will be administered. The parent and clinician will also be asked to rate their perceived itch severity on a full-cartoon version of the ItchyQuant. The ItchyQuant is a 10-point numeric rating scale to rate itch severity. The items are scored from 0-10, where 0=no itch and 10= worst imaginable itch. The validity of the ItchyQuant will be assessed by comparing the responses.
ItchyQoL (TotsItchyQoL) test-retest reliability | 1 hour from baseline
  Subjects in the 4-7 year age group will complete the TotsItchyQoL® questionnaire. This questionnaire has a total of 16 items with cartoons accompanying each question. The interviewer will ask the subjects questions to rate how pruritus affected their quality of life (QOL). The test-retest reliability will be assessed by analyzing the recorded responses to assess improvement, no change, or worsening of their pruritus.
ItchyQoL (TotsItchyQoL) test-retest reliability | 6 months
  Subjects in the 4-7 year age group will complete the TotsItchyQoL® questionnaire. This questionnaire has a total of 16 items with cartoons accompanying each question. The interviewer will ask the subjects questions to rate how pruritus affected their quality of life (QOL). The test-retest reliability will be assessed by analyzing the recorded responses to assess improvement, no change, or worsening of their pruritus.
ItchyQoL (KidsItchyQoL) test-retest reliability | 7 days
  Subjects in the 8-17 year age group will complete the KidsItchyQoL® questionnaire. This is a 27-item questionnaire where the subjects are asked to rate how pruritus affected their quality of life (QOL). The test-retest reliability will be assessed by analyzing the recorded responses to assess improvement, no change, or worsening of their pruritus.
ItchyQoL (KidsItchyQoL) test-retest reliability | 6 months
  Subjects in the 8-17 year age group will complete the KidsItchyQoL® questionnaire. This is a 27-item questionnaire where the subjects are asked to rate how pruritus affected their quality of life (QOL). The test-retest reliability will be assessed by analyzing the recorded responses to assess improvement, no change, or worsening of their pruritus.
ItchyQoL (TotsItchyQoL) validity | 1 hour from baseline
  Subjects in the 4-7 year age group will complete the TotsItchyQoL® questionnaire. There are a total of 16 items with cartoons accompanying each question. The subjects will be asked to rate the severity of their pruritus and the responses will be recorded. Each response will be scored and the scores will be compared across pruritus severity; mild,moderate or severe; to assess the validity of the questionnaire.
ItchyQoL (TotsItchyQoL) validity | 6 months
  Subjects in the 4-7 year age group will complete the TotsItchyQoL® questionnaire. There are a total of 16 items with cartoons accompanying each question. The subjects will be asked to rate the severity of their pruritus and the responses will be recorded. Each response will be scored and the scores will be compared across pruritus severity; mild,moderate or severe; to assess the validity of the questionnaire.
ItchyQoL (KidsItchyQoL) validity | 7 days
  Subjects in the 8-17 year age group will complete the TotsItchyQoL® questionnaire. There are a total of 16 items with cartoons accompanying each question. The subjects will be asked to rate the severity of their pruritus and the responses will be recorded. Each response will be scored and the scores will be compared across pruritus severity; mild,moderate or severe; to assess the validity of the questionnaire.
ItchyQoL (KidsItchyQoL) validity | 6 months
  Subjects in the 8-17 year age group will complete the TotsItchyQoL® questionnaire. There are a total of 16 items with cartoons accompanying each question. The subjects will be asked to rate the severity of their pruritus and the responses will be recorded. Each response will be scored and the scores will be compared across pruritus severity; mild,moderate or severe; to assess the validity of the questionnaire.
Psychometric properties of the ItchyQuant | 1 week
  Age-appropriate ItchyQuant will be administered as follows; subjects 4-5 years will use the modified 3-point ItchyQuant, for subjects 6-7 years, the 3-point and 5-point ItchyQuant and for ages 8 and older, the traditional non-cartoon version of the numeric rating scale (NRS) will be administered. The parent and clinician will also be asked to rate their perceived itch severity on a full-cartoon version of the ItchyQuant. The ItchyQuant is a 10-point numeric rating scale to rate itch severity. The items are scored from 0-10, where 0=no itch and 10= worst imaginable itch. The validity of the ItchyQuant will be assessed by comparing the responses.
Psychometric properties of the ItchyQuant | 2 weeks
  Age-appropriate ItchyQuant will be administered as follows; subjects 4-5 years will use the modified 3-point ItchyQuant, for subjects 6-7 years, the 3-point and 5-point ItchyQuant and for ages 8 and older, the traditional non-cartoon version of the numeric rating scale (NRS) will be administered. The parent and clinician will also be asked to rate their perceived itch severity on a full-cartoon version of the ItchyQuant. The ItchyQuant is a 10-point numeric rating scale to rate itch severity. The items are scored from 0-10, where 0=no itch and 10= worst imaginable itch. The validity of the ItchyQuant will be assessed by comparing the responses.

SECONDARY OUTCOMES:
Feasibility of harnessing an electronic platform as assessed by researcher judgement | 1 year from baseline
  The feasibility of an electronic platform for instruments such that mobile technology (i.e., tablets and smartphones) can be utilized in the field to capture the data will be assessed by the researchers. This electronic platform will be able to store and download the data both in summary format (total scores) as well as item level format, capture data across multiple time points, and deposit data into a variety of queryable databases such as spreadsheets, electronic data capture systems.
Prevalence of ADHD symptoms | Baseline
  The prevalence of symptoms of Attention Deficit Hyperactivity Disorder (ADHD) will be assessed by the ADHD screening questionnaire.This consists of an 18-item scale and each item is scored on a 0 to 3 scale, with 0= never or rarely; 1=mild (sometimes), 2=moderate (often); 3=severe (very often). The total score is computed as the sum of the scores on each item. Higher scores indicate increased severity of symptoms.
Prevalence of ADHD symptoms | 2 weeks
  The prevalence of symptoms of Attention Deficit Hyperactivity Disorder (ADHD) will be assessed by the ADHD screening questionnaire.This consists of an 18-item scale and each item is scored on a 0 to 3 scale, with 0= never or rarely; 1=mild (sometimes), 2=moderate (often); 3=severe (very often). The total score is computed as the sum of the scores on each item. Higher scores indicate increased severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Suephy Chen, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States